CLINICAL TRIAL: NCT03213067
Title: Can Metagenomic and Metadata be Combined Using Bioinformatics and Computational Biology Methods to Personalise Patient Treatment.
Brief Title: Mitochondrial and Microbiota Relationship
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — DNA will be extracted from stool samples and the 16S rRNA gene (V4 region) will be sequenced. The DNA will then be stored in the Newcastle Mitochondrial Research Biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mitochondrial Disease Patients: * Male and Females >18 years at the time of screening
  * Patients must have proven genetic disease (confirmed by assessment of heteroplasmy in blood and urine samples) of the m.3243 A>G mutation.
  * Capacity to provide informed consent taken before any study related activities.
  * Ability and willingness to adhere to the protocol, including all appointments.
  * Ability to read and converse in English.
- Healthy Control Group: * Male and Females >18 years at the time of screening
  * Capacity to provide informed consent taken before any study related activities.
  * Ability and willingness to adhere to the protocol, including all appointments.
  * Ability to read and converse in English.

SUMMARY:
Gastrointestinal (GI) dysmotility in patients with mitochondrial disease are increasingly recognized and often include dysphagia, abdominal pain, abdominal distention, bacterial overgrowth, constipation, and in severe cases surgery. Although the proposed pathological mechanisms underlying the development of GI dysmotility remain diverse, potential mechanisms include mitochondrial dysfunction of smooth muscle within the GI tract and visceral myopathy. Moreover, bacteria within the GI tract, termed 'gut microbiota' has also been identified as a key contributor towards GI dysmotility.

Aim: The aim of this study is to assess the role that the gut microbiota has on clinical disease expression in patients with mitochondrial disease.

Objectives: This is a feasibility study to assess:

1. How does clinical disease severity impact upon the gut microbiota in mitochondrial patients compared to healthy controls.
2. How diagnostic and therapeutic approaches for mitochondrial disease be improved.

Methods: This is a pilot study and is part of the Newcastle Mitochondrial Research Biobank. Stool samples will be collected from patients with a Mitochondrial Encephalomyopathy Lactic Acidosis and Stroke-like episodes (MELAS) phenotype carrier of the m.3243 A>G mutation (N=20) from the United Kingdom Medical Research Council (MRC) Centre for Mitochondrial Disease Patient Cohort (RES/0211/7552, the largest cohort of mitochondrial patients in the world) and the mitochondrial clinic and age and gender matched healthy controls (N=20). DNA will be extracted from stool samples and the 16S rRNA gene (V4 region) will be sequenced. This data will be analysed using bioinformatics pipelines and computational biology.

Long Term Goal: To generate novel information relating to how the gut microbiota impacts upon clinical disease expression. This information could then be used to build a predictive model designed to optimise diagnosis and therapeutic treatments. This method also holds potential for use as a model for ageing and diseases associated with mitochondria not working properly, such as diabetes, cancer and Parkinson's disease. This research has the potential to reduce costs to the NHS and improve patient care and their quality of life.

DETAILED DESCRIPTION:
Background Mitochondrial diseases are an important group of inherited neurometabolic disorders that invariably exhibit multi-organ involvement, are relentlessly progressive, and result in significant morbidity and mortality. They may manifest as discrete clinical syndromes such as mitochondrial encephalomyopathy, lactic acidosis, and stroke like episodes (MELAS), chronic and progressive external ophthalmoplegia (CPEO), and maternally inherited deafness and diabetes (MIDD), or more commonly with a wide overlapping spectrum of clinical features, including hypertrophic cardiomyopathy and gastrointestinal (GI) dysmotility. Symptoms arising from gastrointestinal (GI) dysmotility in patients with mitochondrial disease are increasingly recognized and often include dysphagia, abdominal pain, abdominal distention, bacterial overgrowth, constipation, and in severe cases, intestinal pseudo obstruction mimicking an acute surgical abdomen. The high incidence of this was recently confirmed when we surveyed 86 mitochondrial patients about GI symptoms. Sixty five percent of patients experienced GI dysmotility symptoms, including constipation, early satiety, abdominal pain and abdominal distension (under preparation for publication). Although the proposed pathological mechanisms underlying the development of GI dysmotility remain diverse, potential mechanisms include mitochondrial dysfunction of smooth muscle within the GI tract and visceral myopathy. Moreover, bacteria within the GI tract, termed 'gut microbiota' has also been identified as a key contributor towards GI dysmotility.

Rationale To date, there are few effective treatments for patients with mitochondrial disease and those available are predominantly supportive in nature with no proven treatment efficacy, and poor understanding of the links between the gut microbiota, mitochondrial disease, GI dysmotility and patient health and quality of life. Treatments include various antibiotics and laxatives which are generic and not disease specific. Long term effects of drugs are unknown and the impact these have on the GI tract and gut microbiota in mitochondrial disorders are currently unknown. It is essential to optimise supportive therapeutic strategies and design novel modalities to improve clinical management. Although advances in technology now provide more biological information than ever before, the complexity and volume of data generated exceeds the ability to analyse, interpret and translate this information back into the clinical management, highlighting the need to increase clinical analytical capabilities. The use of bioinformatics and computational biology to combine metagenomics data relating to the gut microbiota and metadata (patient characteristics; phenotype/genotype) is one approach to identify and predict what factors, such as drugs, phenotype and genotype, induce gut microbiota dysbiosis.

Elucidating the complexity and workings of the gut microbiota in mitochondrial disease provides a unique approach and deeper understanding of the biology in general, which is currently lacking in primary mitochondrial disorders. This research will contribute to the gut microbiome field and provide a novel insight into the complex microbe:microbe and microbiota-host interactions. The new insights generated here will provide the foundation for interventional studies aimed at manipulating the gut microbiome and relieving disease burden in patients with mitochondrial disease and potentially diseases associated with mitochondrial dysfunction, such as obesity, diabetes and neuro-degenerative disorders such as dementia and Parkinson's disease.

Objectives

The working hypotheses is that patients with mitochondrial disease experience GI dysmotility, and that the gut microbiota accentuates clinical disease severity. This study aims to provide novel information relating to:

1. How does clinical disease severity impact upon the gut microbiota in mitochondrial patients compared to healthy controls.
2. How diagnostic and therapeutic approaches for mitochondrial disease can be improved.

ELIGIBILITY:
Inclusion Criteria:

Mitochondrial Patients

* Male and Females >18 years at the time of screening
* Patients must have proven genetic disease (confirmed by assessment of heteroplasmy in blood and urine samples) of the m.3243 A>G mutation.
* Capacity to provide informed consent taken before any study related activities.
* Ability and willingness to adhere to the protocol, including all appointments.
* Ability to read and converse in English.

Healthy Controls

* Male and Females >18 years at the time of screening
* Capacity to provide informed consent taken before any study related activities.
* Ability and willingness to adhere to the protocol, including all appointments.
* Ability to read and converse in English.

Exclusion Criteria:

* Previous history of contraindicated conditions including stroke, brain lesion(s) or tumour.
* Abnormal clinical results as determined by physician.
* Patient without capacity to provide informed consent.
* Patient's unwillingness to adhere to the protocol, including all appointments.
* Language barriers preventing patients from reading and conversing in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mitochondrial diseases are an important group of inherited neurometabolic disorders that invariably exhibit multi-organ involvement, are relentlessly progressive, and result in significant morbidity and mortality. They may manifest as discrete clinical syndromes such as mitochondrial encephalomyopathy, lactic acidosis, and stroke like episodes (MELAS), chronic and progressive external ophthalmoplegia (CPEO), and maternally inherited deafness and diabetes (MIDD), or more commonly with a wide overlapping spectrum of clinical features, including hypertrophic cardiomyopathy and gastrointestinal (GI) dysmotility (Gorman et al., 2016; Taylor & Turnbull, 2005).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
16S rRNA gene | 6 months
  DNA will be extracted from stool samples and the 16S rRNA gene (V4 region) will be sequenced.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Gorman, MD, Principal Investigator — Consultant Neurologist and Clinical Senior Lecturer
Locations (1):
- Grainne Gorman, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No